CLINICAL TRIAL: NCT04432454
Title: An Open-label, Multicenter Study Evaluating the Safety of Lasofoxifene in Combination With Abemaciclib for the Treatment of Pre- and Postmenopausal Women With Locally Advanced or Metastatic ER+/HER2- Breast Cancer and Have an ESR1 Mutation ( ELAINEII )
Brief Title: Evaluation of Lasofoxifene Combined With Abemaciclib in Advanced or Metastatic ER+/HER2- Breast Cancer With an ESR1 Mutation
Acronym: ELAINEII
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sermonix Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMX 20-001
Record Dates: First submitted 2020-06-04; First posted 2020-06-16 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Lasofoxifene; abemaciclib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Women who have locally advanced or metastatic ER+/HER2- breast cancer and disease progression on first and/or 2nd lines of hormonal treatment for metastatic disease and have an ESR1 mutation
  Interventions: Drug: Lasofoxifene and abemaciclib (VERZENIO (R)).

INTERVENTIONS:
Drug: Lasofoxifene and abemaciclib (VERZENIO (R)). — Lasofoxifene 5 mg given once a day orally and abemaciclib 150 mg given twice a day orally.

SUMMARY:
This is an open-label, multicenter, single-arm safety study evaluating the safety and tolerability of the lasofoxifene and abemaciclib combination for the treatment of pre- and postmenopausal women with locally advanced or metastatic ER+/HER2- breast cancer who have disease progression on first and/or 2nd lines of hormonal treatment for metastatic disease and have an ESR1 mutation.

ELIGIBILITY:
Inclusion Criteria:

1. Pre- or postmenopausal.

   Postmenopausal women are defined as:
   1. ≥ 60 years of age with no vaginal bleeding over the prior year, or
   2. < 60 years with "premature menopause" or "premature ovarian failure" manifest itself with secondary amenorrhea for at least 1 year and follicle stimulating hormone (FSH) and estradiol levels in the postmenopausal range according to institutional standards, or
   3. surgical menopause with bilateral oophorectomy. Note: Premenopausal women who meet all of the other entry criteria must be maintained on ovarian suppression (such as Lupron) during the study and subjects counseled to use appropriate contraception to prevent pregnancy.
2. If possible, a biopsy of metastatic breast cancer tissue should be obtained to provide histological or cytological confirmation of ER+/HER2- disease as assessed by a local laboratory, according to American Society of Clinical Oncology/College of American Pathologists guidelines, using slides, paraffin blocks, or paraffin samples. If a biopsy is not possible, the ER and HER2 status from the tissue obtained at the time of the original diagnosis must confirm that the subject is ER+ and HER2-.
3. Locally advanced and/or metastatic breast cancer with radiological or clinical evidence of progression on the first or 2nd lines of hormonal therapy for metastatic disease. Progression may have occurred on no more than 2 of the following endocrine treatments for metastatic breast cancer: an aromatase inhibitor (AI) and/or fulvestrant either as monotherapy or in combination with any commercially approved CDKi; and/or the combination of fulvestrant and everolimus; and/or the combination of fulvestrant and alpelisib; and/or tamoxifen; and/or the combination of exemestane/everolimus. (Note: before starting study treatment, subjects should have stopped any CDKi for at least 21 days)
4. Subjects must have had no evidence of progression for at least 6 months during their first hormonal treatment for advanced breast cancer.
5. At least one or more of the following ESR1 point mutations as assessed in cell-free circulating tumor DNA (ctDNA) obtained from a blood or tissue sample: Y537S, Y537C, D538G, E380Q, S463P, V534E, P535H, L536H, L536P, L536R, L536Q, or Y537N. Note: the Sponsor's blood ctDNA assay must be used but tissue sequencing (if done) may be done by a validated commercial laboratory.

   Note: A positive ESR1 mutation in tissue or ctDNA using a validated commercial assay if done prior or at the time of disease progression is acceptable to meet this entry criteria. However, blood for ctDNA must still be obtained for genomic analyses using the sponsor's ctDNA assay.
6. Locally advanced or metastatic breast cancer with either measurable (according to RECIST 1.1) or non-measurable lesions.
7. Subjects may have received one cytotoxic chemotherapy regimen for metastatic disease as well as those who received one cytotoxic chemotherapy regimen in the neo-adjuvant or adjuvant setting prior to entry into the trial can be enrolled but must be free of all chemotherapy acute toxicity excluding alopecia and Grade 2 peripheral neuropathy before study entry. A washout period of at least 21 days is required between last chemotherapy dose and entry into the study.
8. Stable breast cancer metastasis to the brain is allowed as long as the subject has received radiotherapy and not demonstrated any evidence of brain metastasis progression for at least 3 months after the completion of radiotherapy.
9. ECOG performance score of 0 or 1.
10. Adequate organ function as shown by:

    1. absolute neutrophil count (ANC) ≥ 1,500 cells/mm3
    2. platelet count ≥ 100,000 cells/mm3
    3. hemoglobin ≥ 8.0 g/dl
    4. ALT and AST levels ≤ 3 upper limit of normal (ULN) or ≤ 5 in the presence of liver metastasis
    5. total serum bilirubin ≤ 1.5 X ULN (≤ 3 X ULN for subjects known to have Gilbert Syndrome)
    6. alkaline phosphatase level ≤ 3 ULN
    7. creatinine clearance of 40 ml/min or greater as calculated by the Cockcroft-Gault formula
    8. International normalized ratio (INR) and activated partial thromboplastin (aPTT) < 2.0 X ULN
11. Able to swallow tablets.
12. Able to understand and voluntarily sign a written informed consent before any screening procedures.

Exclusion Criteria:

1. Lymphangitic carcinomatosis involving the lung.
2. Visceral crisis in need of cytotoxic chemotherapy as assessed by the investigator.
3. Radiotherapy within 30 days prior to entry into the study except in case of localized radiotherapy for analgesic purposes or for lytic lesions at risk of fracture, which can then be completed within 7 days prior to entry into the study. Subjects must have recovered from radiotherapy toxicities prior to entry into the study.
4. Subjects with known inactivating RB1 mutations or deletions (Screening for RB1 mutation is not required for entry).
5. History of long QTC syndrome or a QTC of > 480 msec.
6. History of a pulmonary embolus (PE) or deep vein thrombosis (DVT) within the last 6 months or any known thrombophilia. Subjects stable on anti-coagulants for maintenance are eligible as long as the DVT and/or PE occurred > 6 months prior to enrollment and there is no evidence for active thrombosis. The use of low-dose ASA is permitted.
7. Subjects on concomitant strong CYP3A4 inhibitors such as clarithromycin, telithromycin, nefazodone, itraconazole, ketoconazole, atazanavir, darunavir, indinavir, lopinavir, nelfinavir, ritonavir, saquinavir, tipranavir.
8. Subjects on strong and moderate CYP3A4 inducers such as amprenavir, barbiturates, carbamazepine, clotrimazole, dexamethasone, efavirenz, ethosuximide, griseofulvin, modafinil, nevirapine, oxcarbazepine, phenobarbital, phenytoin, chronic prednisone treatment, primidone, rifabutin, rifampin, rifapentine, ritonavir, topiramate.
9. Any significant co-morbidity that would impact the study or the subject's safety. Since CDKi have reported the occurrence of interstitial lung disease (ILD), subjects with a history of ILD and those with severe dyspnea at rest or requiring oxygen therapy should not enter the study
10. Subject has an active systemic bacterial or fungal infection (requiring intravenous [IV] antibiotics at the time of initiating study treatment).
11. History of a positive human immunodeficiency virus (HIV) or hepatitis B virus (HBV) test. Screening is not required for enrollment.
12. Subjects with hepatitis C virus (HCV) at Screening who still have a viral load. Subjects previously treated and achieved a HCV cure (no viral load) can be entered into the study
13. History of malignancy within the past 5 years (excluding breast cancer), except basal cell or squamous cell carcinoma of the skin curatively treated by surgery, or early-stage cervical cancer.
14. Positive serum pregnancy test (only if premenopausal).
15. History of non-compliance to medical regimens.
16. Unwilling or unable to comply with the protocol.
17. Current participation in any clinical research trial involving an investigational drug or device within the last 30 days.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 29 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2025-01-28 (Actual); Study Completion 2025-01-28 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of the combination of lasofoxifene and abemaciclib as measured by number of adverse events (AEs), severity of AEs and mortality due to AEs at every scheduled visit. | All subjects enrolled in the study will be treated until documented disease progression or until withdrawal for any reason. Safety and tolerability will be assessed from enrollment up to 24 months.
  AEs will be assessed by the Common Terminology Criteria for Adverse Events (CTCAE) version 5.

SECONDARY OUTCOMES:
Progression free survival (PFS) | Up to 24 months
  PFS is defined as the time from the date of entry into the study to the earliest date of first documented progression or death due to any cause.
Clinical benefit rate (CBR) | 24 weeks or longer
Objective response rate (ORR) | All subjects enrolled in the study will be treated until documented disease progression or until withdrawal for any reason. ORR will be assessed up to 24 months.
Duration of response (DoR) | DoR will be assessed up to 24 months.
  DoR is from the date of first documented response (CR or PR) to the date of first documented progression of disease or death due to any cause.
Time to response | Time to response will be assessed up to 24 months.
  From the date of entry into the study to the date of first documented response (CR or PR).
Steady-state pharmacokinetics (PK) sampling for lasofoxifene and abemaciclib concentrations as well as abemaciclib's 3 major metabolites | Baseline and pre-dose at every visit starting at Visit 0 (Day 1) through Visit 4 (Week 8) and at the Final/ET visit if this occurred prior to Week 8

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - University of Alabama at Birmingham (UAB) - Comprehensive Cancer Center, Birmingham, Alabama
  - Yuma Regional Medical Center, Yuma, Arizona
  - Compassionate Cancer Care Med Group - Clinic Aid USA - Fountain Valley, Fountain Valley, California
  - St. Joseph Health, Santa Rosa, California
  - Mayo Jacksonville, Jacksonville, Florida
  - Illinois Cancer Care, Peoria, Illinois
  - Beacon Health System Memorial Regional Cancer Center, South Bend, Indiana
  - Mayo Clinic Rochester, Rochester, Minnesota
  - New Jersey Cancer Care, PA, Belleville, New Jersey
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mary Crowley Cancer Research, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Oncology Consultants, P.A., Houston, Texas
  - Hematology Oncology Associates of Fredericksburg, Fredericksburg, Virginia
  - Northwest Medical Specialists, PLLC (NWMS), Tacoma, Washington

REFERENCES:
- [Derived] Damodaran S, O'Sullivan CC, Elkhanany A, Anderson IC, Barve M, Blau S, Cherian MA, Peguero JA, Goetz MP, Plourde PV, Portman DJ, Moore HCF. Open-label, phase II, multicenter study of lasofoxifene plus abemaciclib for treating women with metastatic ER+/HER2- breast cancer and an ESR1 mutation after disease progression on prior therapies: ELAINE 2. Ann Oncol. 2023 Dec;34(12):1131-1140. doi: 10.1016/j.annonc.2023.09.3103. PMID 38072513
- [Derived] Blau S, Peguero JA, Moore HCF, Anderson IC, Barve MA, Cherian MA, Elkhanany A, O'Sullivan CC, Moreno-Aspitia A, Plourde P, Gleich LL, Riesen K, Ezzati R, Degele M, Shulman M, Stempf SD, Sachse L, Iyer AA, Damodaran S, Cooney MM. Operational Metrics for the ELAINE 2 Study Combining a Traditional Approach With a Just-in-TIME Model. JCO Clin Cancer Inform. 2023 Jun;7:e2200164. doi: 10.1200/CCI.22.00164. PMID 37352479